CLINICAL TRIAL: NCT06938074
Title: Imaging and Treatment Planning for Cardiac Radioablation
Acronym: ITPCR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stewart Gaede (Other)
Responsible Party: Sponsor-Investigator, Stewart Gaede, Chief Medical Physicist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 126882
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Ventricular Tachycardia, Monomorphic; Ventricular Tachycardia (V-Tach); Ischemia, Myocardial
Keywords: Cardiac radioablation; Stereotactic arrhythmia radioablation; Ischemic fibrosis; Late iodine enhancement CT; CT perfusion; Late gadolinium enhanced MRI
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Ischemia | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT and MRI (Experimental): All participants will undergo both CT imaging and MRI imaging to identify areas of ischemic scar. Treatment plans will be created based on CT scans, using various treatment delivery and motion management techniques.
  Interventions: Diagnostic Test: CT and MRI

INTERVENTIONS:
Diagnostic Test: CT and MRI — All participants will undergo both CT imaging and MRI imaging to identify areas of ischemic scar. Treatment plans will be created based on CT scans, for all participants using various treatment delivery and motion management techniques.

SUMMARY:
Cardiac radioablation is a new treatment for ventricular tachycardia (VT), which uses beams of radiation to treat heart scar that causes VT. To identify the scar areas, magnetic resonance imaging (MRI) and computed tomography (CT) imaging are often used. These are both types of medical imaging that allow clinicians to examine scar area without having to do invasive surgery.

Researchers have developed new heart imaging protocols using both MRI and CT. Their MRI protocol method can now spot both dense and scattered scar tissue. The CT protocol combines multiple different types of scans into a single appointment and uses a special scanner that captures the motion of the heart. For this study, patients will undergo CT and MRI imaging according to these new imaging protocols.

With this study, researchers aim to show that these new imaging protocols can be undergone by patients with ventricular tachycardia and can be used to identify scar. Researchers will also use these scans to make radiation treatment plans to identify which types of treatment can be delivered safely to patients.

ELIGIBILITY:
Inclusion Criteria

* Ischemic cardiomyopathy with monomorphic VT
* Referred by cardiologists
* 18 years of age or older Exclusion Criteria
* • Polymorphic ventricular tachycardia
* Ventricular fibrillation
* Pregnant or breastfeeding or planning to become pregnant or breastfeed during the study
* Estimated glomerular filtration rate ≤ 30 mL/min/1.73m2
* Previous allergic reaction to CT contrast agent Note that participants with contraindications for MRI can still be enrolled in this study but will not undergo MRI parts of this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Agreement among cardiologists for target regions, assessed by an inter- and intra-observer variability study using similarity metrics such as the Dice coefficient and Hausdorff distance. | 6 months after conclusion of study
  Imaging protocols will be delivered to participants. Targets will be delineated by experts. Agreement between experts will be assessed..
Adherence of treatment plans to dose constraints and deliverability of treatment plans. | 6 months after conclusion of study
  Treatment plans will be created using various motion management and radiation treatment delivery strategies. Adherence of treatment plans to dose constraints will be assessed by comparing treatment plans to institutional dose constraints. Beam deliverability will be assessed by delivering the treatment plan to a static phantom and comparing the deposited dose to the expected dose. Treatment deliverability, as it relates to motion management, will be assessed by delivering the treatment plan to a moving phantom and comparing the deposited dose to the expected dose.

SECONDARY OUTCOMES:
Agreement between CT/MRI areas of interest (scar), assessed using similarity metrics such as the Dice coefficient and Hausdorff distance. | 6 months after conclusion of study

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre Research Inc, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No